CLINICAL TRIAL: NCT06110559
Title: Use of tDCS (Transcranial Direct Current Stimulation) Applied to the Orbitofrontal Cortex to Improve Risky Decision-making in a Clinical Population: a Proof-of-concept Study
Brief Title: Use of tDCS Applied to the Orbitofrontal Cortex to Improve Risky Decision-making in a Clinical Population
Acronym: tDCSDeMOStim
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D20-P041
Record Dates: First submitted 2023-10-19; First posted 2023-10-31 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Mood Disorders; Depression; Suicide
Keywords: Endophenotype; Transcranial Direct Current Stimulation; Cognition
MeSH Terms: conditions — Mood Disorders; Depression; Suicide

STUDY DESIGN:
Intervention Model Description: Prospective monocentric interventional randomised controlled trial vs placebo (sham tDCS) in 2 parallel groups.
  An interim analysis focusing on the primary objective will be performed when at least 50% of the total expected sample has completed the study.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients and the outcome assessor are blinded to the type of treatment received.
  Each patient, at the end of the study, will be asked to guess whether the treatment received was active or sham.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS active comparator (Experimental): Active transcranial Direct Current Stimulation (tDCS): Stimulation of 1.5 mA for 30 minutes.
  Interventions: Device: Active transcranial direct current stimulation (tDCS)
- tDCS sham comparator (Sham Comparator): Sham transcranial Direct Current Stimulation (tDCS): Effective stimulation of 1.5 mA for 30 seconds, then the current is switched off. The complete session lasts 30 minutes, with 29 minutes and 30 seconds without stimulation.
  Interventions: Device: Sham transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: Active transcranial direct current stimulation (tDCS) — Description of the tDCS session:
  * Placement of conductive electrodes, attached to the scalp. The electrodes are placed in individual sponge cases moistened with a saline solution. A sponge towel is placed on the patient's shoulders to prevent any clothing from becoming damp. The electrodes are held in place by a dedicated net.
  * The anode is placed in the left supraorbital region (site Fp1 EEG 10/20 system). The cathode was placed in the right supraorbital region (site Fp2 EEG 10/20 system).
  * Patients received 1.5 mA stimulation for 30 minutes.
  Arms: tDCS active comparator
Device: Sham transcranial direct current stimulation (tDCS) — Description of the tDCS session:
  * Placement of conductive electrodes, attached to the scalp. The electrodes are placed in individual sponge cases moistened with a saline solution. A sponge towel is placed on the patient's shoulders to prevent any clothing from becoming damp. The electrodes are held in place by a dedicated net.
  * The anode is placed in the left supraorbital region (site Fp1 EEG 10/20 system). The cathode was placed in the right supraorbital region (site Fp2 EEG 10/20 system).
  * Patients received effective stimulation of 1.5 mA for 30 seconds, after which the current was switched off. The entire session lasted 30 minutes, with 29 minutes and 30 seconds without stimulation.
  Arms: tDCS sham comparator

SUMMARY:
Decision-making is a complex cognitive function that has been the subject of extensive scientific research in the fields of cognitive and computational neuroscience. It relies on a cerebral network that encompasses cortico-subcortical pathways. The orbitofrontal cortex (OFC) plays a significant role in decision-making by assigning values to guide choices. Risky decision-making is observed in several psychiatric pathologies, including depression and bipolar disorder, and it may constitute an endophenotype of suicide. In the project presented here, we propose to use transcranial direct current stimulation (tDCS) to target decision-making in patients suffering from mood disorders.

DETAILED DESCRIPTION:
The primary objective is to assess the ability of tDCS applied to the orbitofrontal cortex to improve decision-making, as measured by the Iowa Gambling Task, compared to a placebo stimulation in patients suffering from mood disorders.

The secondary objectives are as follows:

* To assess whether the evolution of decision-making under tDCS stimulation is independent of emotional changes (sadness, anxiety).
* To evaluate if tDCS stimulation of the orbitofrontal cortex improves motor inhibition, assessed using the D2-test, compared to a placebo stimulation.
* To determine if tDCS stimulation of the orbitofrontal cortex reduces sensitivity to interference, assessed with the Stroop test, compared to a placebo stimulation.
* To evaluate if tDCS stimulation of the orbitofrontal cortex enhances cognitive inhibition, measured by the Go-no go test, compared to a placebo stimulation.

This is a prospective monocentric interventional randomised controlled trial with two parallel groups, one receiving active treatment with tDCS and the other receiving a placebo (sham tDCS). The randomization will be performed in variable-sized blocks and will be stratified based on the current mood state (current depression versus current euthymia). It is a single-blind study where the patients and the outcome assessor are blinded to the type of treatment received.

Recruitment will take place at "la Clinique des Maladies Mentales et de l'Encéphale de l'Hôpital Sainte-Anne" and will involve hospitalized patients as well as those in outpatient care. Pre-inclusion visit involve patient selection, verification of inclusion criteria, and the provision of information documents. Inclusion visit occur at least one day later, lasting for three hours. It involves the verification of both inclusion and exclusion criteria, obtaining informed consent, randomization, collecting socio-medical-demographic data, and conducting psychometric and neuropsychological assessments. Stimulation visit, also scheduled at least one day later and lasting three hours, encompass the measurement of primary and secondary evaluation criteria immediately before and after tDCS stimulation. A group guessing test concludes the study.

An interim analysis is planned, and an Independent Data Monitoring Committee (IDMC) will be established to oversee the data.

ELIGIBILITY:
Inclusion Criteria:

* Patients under consideration should either be receiving outpatient or inpatient care.
* Patients must be between the ages of 18 and 65, inclusive.
* According to DSM-5 criteria, patients should be diagnosed with either unipolar or bipolar depressive disorder. This includes individuals currently experiencing a characterized depressive episode with mild to moderate intensity, those in partial remission, or those in full remission.
* Patients must have provided informed consent.
* Patients should be enrolled in a social security plan.

Exclusion Criteria:

* Patient unwilling to participate in the research.
* Non-French-speaking individuals.
* Individuals deprived of liberty by judicial or administrative decision, such as those under guardianship or curatorship or involuntarily hospitalized.
* Pregnant or breastfeeding women.
* Current hypomanic or manic episode as per DSM-5 criteria due to motor agitation issues.
* Ongoing electroconvulsive therapy (ECT) treatment or within the last 6 months.
* Patients with active implantable medical devices.
* Epilepsy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2021-04-16 (Actual); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
The study aims to assess the effectiveness of tDCS applied to the orbitofrontal cortex in enhancing decision-making abilities, as measured by the Iowa Gambling Task, when compared to placebo stimulation in patients with mood disorders. | Day 1 (end of study)
  The primary outcome measure is the net score on the Iowa Gambling Task over 100 selections. This score represents the difference between the number of selections from low-risk and long-term advantageous decks and the number of selections from high-risk and long-term disadvantageous decks during 100 selections. This score ranges from -100 to 100, and the lower the score, the riskier the decision-making. This measurement will be taken immediately before and after tDCS stimulation.

SECONDARY OUTCOMES:
To assess whether the change in decision-making under tDCS stimulation is independent of emotional changes (sadness). | Day 1 (end of study)
  PANAS : Positive and Negative Affect Schedule. Positive Affect Score range from 10 - 50, with higher scores representing higher levels of positive affect Negative Affect Score range from 10 - 50, with lower scores representing lower levels of negative affect.
To assess whether the change in decision-making under tDCS stimulation is independent (STAI:State-Trait Anxiety Inventory) | Day 1 (end of study)
  STAI score range from 20 to 80. STAI scores are commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80).
  These measurements will be taken immediately before and after tDCS stimulation.
To assess whether tDCS stimulation of the OFC improves motor inhibition compared to placebo stimulation (Sustained-Attention test: d2-test) | Day 1 (end of study)
  d2-test: the test taker is required to scan the lines and cross out all occurrences of the letter 'd' with two dashes while ignoring all other characters. During the test, the subject must delete as many 'd2' as possible in 20 seconds per line (there are 14 lines on the sheet).
  This measurement will be taken immediately before and after tDCS stimulation.
To assess whether tDCS stimulation of the OFC improves reduces susceptibility to interference compared to placebo stimulation. | Day 1 (end of study)
  Emotional stroop task : Difference in reaction time. The higher the score, the greater the susceptibility to interference. This measurement will be taken immediately before and after tDCS stimulation.
To assess whether tDCS stimulation of the OFC improves cognitive inhibition compared to placebo stimulation. | Day 1 (end of study)
  Go-no go task : Commission error rate. The lower the score, the more effective cognitive inhibition is. This measurement will be taken immediately before and after tDCS stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Michel DANON, MD, Principal Investigator — GHU Paris Pyschiatrie & Neurosciences
Locations (1):
- GHU Paris Psychiatrie et Neurosciences - Hôpital Sainte-Anne - CMME, Paris, France